CLINICAL TRIAL: NCT00949598
Title: Randomized Double-blind Study to Compare Two Neo-adjuvant Treatments: an Anti-aromatase vs SERM for Postmenopausal Women With ER+ Breast Adenocarcinoma: Effect on Intermediate Predictive Biological Response to Treatment.
Brief Title: Letrozole or Tamoxifen Citrate in Treating Older Postmenopausal Women Undergoing Surgery for Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CDR0000638373
Record Dates: First submitted 2009-07-29; First posted 2009-07-30 (Estimated); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Breast Cancer
Keywords: estrogen receptor-positive breast cancer; stage IA breast cancer; stage IB breast cancer; stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole; Tamoxifen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Experimental): Patients receive oral letrozole once daily for 16 weeks.
  Interventions: Drug: letrozole
- Arm II (Experimental): Patients receive oral tamoxifen citrate once daily for 16 weeks.
  Interventions: Drug: tamoxifen citrate

INTERVENTIONS:
Drug: letrozole — Given orally
  Arms: Arm I
Drug: tamoxifen citrate — Given orally
  Arms: Arm II

SUMMARY:
RATIONALE: Estrogen can cause the growth of breast cancer cells. Hormone therapy using letrozole may fight breast cancer by blocking the uptake of estrogen. Tamoxifen citrate may fight breast cancer by blocking the use of estrogen by the tumor cells. It is not yet known whether letrozole or tamoxifen citrate is more effective when given before surgery in treating older women with breast cancer.

PURPOSE: This randomized phase III trial is studying letrozole to see how well it works compared with tamoxifen citrate in treating older postmenopausal women undergoing surgery for breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Investigate the changes in Ki67 and PCNA in postmenopausal women with estrogen receptor-positive (ER+) breast cancer after 4 months of treatment with letrozole vs tamoxifen citrate.

Secondary

* Compare the response after 4 months of therapy.
* Define the resistant forms of cancer in patients treated with these regimens.
* Define the molecular signature predictive of sensitivity or resistance to ER+ breast adenocarcinoma by gene and serum protein profiling.
* Search for serum protein profiles predictive of recurrence-free interval.

OUTLINE: Patients are randomized into 1 of 2 intervention arms.

* Arm I: Patients receive oral letrozole once daily for 16 weeks.
* Arm II: Patients receive oral tamoxifen citrate once daily for 16 weeks. Patients in both arms then undergo surgery.

Blood and tumor tissue samples are collected at baseline and after completion of neoadjuvant therapy for changes in Ki67 and PCNA and serum protein profiling analysis.

After completion of study therapy, patients are followed up every 6 months for 3 years, and then once a year for 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed invasive breast adenocarcinoma

  * Clinically T2 tumor and/or > 1 cm by echography
  * Estrogen receptor (ER)-positive and > 10% of the tumor cells positive

    * No ER-negative disease
* No prior breast cancer
* No metastatic or inflammatory breast adenocarcinoma

PATIENT CHARACTERISTICS:

* Postmenopausal
* No cardiac function that could contraindicate surgery or medical treatment (e.g., radiotherapy and/or chemotherapy)
* No prior malignancies within the past 5 years except for nonmelanoma skin cancer or carcinoma in situ of the cervix
* No mental incapacitation that would preclude consent
* No contraindication to tamoxifen citrate or letrozole

PRIOR CONCURRENT THERAPY:

* More than 8 days since prior hormone-replacement therapy or other treatment (i.e., phytoestrogen) for menopause
* No concurrent therapy that would modify the expression of the genes regulated by estrogen
* No concurrent participation in another clinical study

Ages: 65 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 177 (Actual)
Dates: Start 2008-12; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Changes in Ki67 and PCNA after 4 months of treatment with letrozole vs tamoxifen citrate | up to 24 months

SECONDARY OUTCOMES:
Molecular signature predictive of sensitivity or resistance to estrogen receptor-positive breast adenocarcinoma | up to 24 months
Survival rate | up to 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Rouanet, MD, PhD, Principal Investigator — Institut du Cancer de Montpellier - Val d'Aurelle
Locations (1):
- Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier, France